CLINICAL TRIAL: NCT01517958
Title: The Use of Lung Ultrasound to Diagnose RDS vs. TTN in Neonates Greater Than or Equal to 28 Weeks Gestation
Brief Title: Lung Ultrasound to Diagnose Transient Tachypnea of the Newborn (TTN) Versus Respiratory Distress Syndrome (RDS) in Neonates
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 11-0598; IF#1289354
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Transient Tachypnea of the Newborn; TTN; Respiratory Distress Syndrome; RDS
Keywords: Transient tachypnea of the newborn; Respiratory Distress Syndrome; Lung Ultrasound; Neonates
MeSH Terms: conditions — Transient Tachypnea of the Newborn; Respiratory Distress Syndrome | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Respiratory Distress Group: Neonates 28 weeks GA or greater with respiratory distress
  Interventions: Other: Respiratory Distress Group
- Control Group: Neonates 28 weeks GA or greater without respiratory distress.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Respiratory Distress Group — Diagnostic lung ultrasound.
  Other Names: Diagnostic lung ultrasound.
  Groups: Respiratory Distress Group
Other: Control Group — Lung ultrasound
  Groups: Control Group

SUMMARY:
The investigators hypothesize that ultrasonography of the newborn lung can be used as an effective diagnostic tool in neonates ≥ 28 weeks gestation with early symptoms of respiratory distress.

DETAILED DESCRIPTION:
Respiratory distress is a common reason for admission to the neonatal intensive care unit (NICU) for both preterm and full term newborns. TTN and RDS are the two most common diagnoses associated with respiratory distress. Due to their similar clinical presentations, it is often difficult to differentiate the two diseases clinically. Currently chest radiography is used to differentiate between TTN and RDS, however, radiographic findings are not always definitively diagnostic.

In preliminary studies, lung ultrasonography has been shown to be a useful tool in diagnosing both TTN and RDS. However, no one has looked at the use of lung ultrasonography in differentiating TTN from RDS in the neonatal population. We propose to do so in this study.

Patients will be enrolled from neonatal admissions to the NICU with respiratory distress. Lung ultrasound will be performed on all enrolled subjects, looking for specific findings suggestive of either TTN or RDS. Data will be collected on gestational age, physical exam findings and level of respiratory support. Diagnoses will be recorded based on ultrasound findings. Accuracy of lung ultrasound diagnosis will be compared to that using radiographic chest radiography findings to evaluate if lung ultrasound is equivalent, or better than chest radiography in order to diagnose TTN versus RDS in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≥ 28 weeks
* symptoms of respiratory distress defined as:
* tachypnea (respiratory rate > 60 breaths per minute)
* FiO2 requirement >21%
* intercostal/subcostal retractions
* grunting and/or nasal flaring
* If clinically warranted, a chest x-ray will be done as part of the workup for respiratory distress; these patients with CXR will be included in the study.
* Inclusion criteria for the control group will be gestational age ≥ 28 weeks with no symptoms of respiratory distress (defined above).

Exclusion Criteria:

* neonates with prenatally diagnosed structural cardiac disease
* major multiple congenital anomalies
* other causes of respiratory distress that are not RDS or TTN (e.g. pneumothorax, CCAM or pneumonia).

Min Age: 28 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Neonatal patients admitted to Mount Sinai NICU of gestational age greater than or equal to 28 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
lung ultrasound | within first 24 hours of life.
  The primary endpoint is to determine whether lung ultrasound is comparable or superior to chest radiography: (1) in making the diagnosis of RDS and TTN and (2) in differentiating between RDS and TTN.
  Disease-specific lung ultrasound findings: (1) Double lung point in TTN and (2) lung white-out in RDS.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Holzman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No